CLINICAL TRIAL: NCT06414096
Title: Use of Pulsatile Intravenous FSH to Mitigate Reprometabolic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23-2564b
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Infertility; Obesity
MeSH Terms: conditions — Infertility; Obesity | interventions — Follicle Stimulating Hormone

STUDY DESIGN:
Intervention Model Description: Examine effects of pulsatile FSH administration as a new method for stimulation in IVF
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Conventional Subcutaneous FSH Dosing (Active Comparator): A daily gonadotropin dose (typically 75-450 IU) will be assigned and adjusted, based on clinical criteria and, if known, past response to hormones. Recombinant human FSH (rhFSH) will be given as a daily subcutaneous injection, as is performed, by patients at home, in routine clinical practice.
  Interventions: Drug: Follicle Stimulating Hormone
- Pulsatile IV FSH Dosing (Experimental): participants will receive the same daily rhFSH dose (based on clinical practice criteria); however, it will be delivered via a portable infusion pump with reservoir (Avocet Infusion Pump, Eitan Medical LTD) that will provide an IV bolus (100-500 µl) every 90 minutes, a frequency that has previously been shown to result in physiologic ovulatory cycles in GnRH deficient women (Martin). The total gonadotropin dose delivered over a 24 hour period will be typically 75-450 IU, assigned based on standard of care clinical criteria (max dose is 900IU per clinical care guidelines). Participants will be provided with a 100mL preloaded reservoir, calibrated to deliver the approved standard of care dosing, in 16 boluses (100-500µl) over 24 hours (q 90min), for 7-12 days. Each 100 ml reservoir has capacity for 200 doses if the volume is 500 µl, which is sufficient for the typical 7- 12-day protocol.
  Interventions: Drug: Follicle Stimulating Hormone

INTERVENTIONS:
Drug: Follicle Stimulating Hormone — Pulsatile FSH administration via a portable pump.
  Other Names: FSH

SUMMARY:
Hypothesis: The investigators hypothesize that pulsatile FSH intravenous administration to women with obesity will correct the Reprometabolic Syndrome (RMS) luteal deficiency phenotype.

Specific Aim: To test the hypothesis that pulsatile IV administration of FSH will rescue the impaired folliculogenesis and relative hypogonadotropic hypogonadism, characteristic of obesity. The investigators will accomplish this by administering a cycle of pulsatile FSH to women with obesity and comparing their hormone output to a cycle using conventional, daily FSH injection at the identical daily dose. The primary outcome will be luteal phase progesterone excretion.

DETAILED DESCRIPTION:
Design: Crossover interventional study. The investigators have selected this design to allow us to compare each woman to herself in consecutive cycles whenever possible.

Methods:

Patient population and protocol: The investigators plan to recruit women with obesity for a proof-of-concept study to demonstrate the potential of this treatment to improve fertility. Before such a treatment would be brought into clinical practice, a more comprehensive program of pre-conceptional care would be desirable to improve the metabolic health of women with obesity and minimize pregnancy complications such as preterm birth and pregnancy related hypertension.

However, that is not the goal of this preliminary study which only seeks to identify reproductive hormone impact.

Consent/Screening Process: A script for screening participants by telephone who inquire in response to advertisements will be used, which will include the required verbal consent language. Participants who are eligible for enrollment will be asked to come to the Clinical and Translational Research Center (CTRC) for an intake examination and qualifying laboratory tests. At this time, informed consent is obtained by the PI, the Professional Research Assistant, or an Institutional review Board (IRB) approved designee, according to the scripted process. The informed consent discussion is always held in a private room that is free of distractions and participants are allowed the opportunity to ask questions and have their questions answered to their satisfaction before signing the informed consent document. Once informed consent has been provided, procedures are performed as outlined in the procedures section.

The investigators will prepare the participants for either a cycle of pulsatile FSH or conventional, daily FSH injection at the identical daily dose of FSH for both conditions. Participants will be randomized to group A, pulsatile FSH and then conventional daily injected FSH, or group B, conventional FSH and then pulsatile FSH, by the study statistician. Participants will not be blinded to treatment. However, the PI and co-investigator, as well as the research assistant who will perform the assays, will not be expected to be involved in direct care of participants during treatment and will therefore be able to remain blinded to treatment assignment.

To control hormone delivery for both conditions (non-pulsatile FSH vs pulsatile FSH), all participants will receive a Gonadotropin Releasing Hormone (GnRH) antagonist during gonadotropin stimulation and up to the day of Human Chorionic Gonadotropin (HCG) trigger to abolish endogenous gonadotropin production. A baseline ultrasound will be performed within 2 days of the onset of menses to assure that no dominant follicles are present on ovarian ultrasound and E2 is <50 pg/ml prior to initiating stimulation, as per usual clinical practice. The remaining protocol will be administered in the second cycle, after a 1-month 'washout' period to avoid the possibility of carryover.

ELIGIBILITY:
Inclusion Criteria:

* • BMI between 30 kg/m2 and 40 kg/m

  * Weight stability, i.e. no continued weight loss of >1lb per week for a minimum of 4 weeks prior to enrollment
  * Normal thyroid stimulating hormone (TSH) and prolactin
  * Anti-Mullerian Hormone (AMH) > 1 ng/ml or < 8 ng/mL
  * Willingness to postpone conception for the first study cycle
  * Involuntary inability to conceive for at least 6 months
  * No clinical diagnosis of polycystic ovarian syndrome (PCOS)
  * Documentation of ovulation with luteal progesterone >6 ng/ml or positive ovulation predictor home testing
  * Regular menstrual cycles 25-40 days in length
  * Male partner (or sperm donor) with adequate sperm (>14 million sperm per ml)
  * Hysterosalpingogram or saline infusion sonography demonstrating at least one patent Fallopian tube and a normal uterine cavity
  * Serum total and free testosterone within the 95% CIearance for women with obesity previously studied in our laboratory.
  * Acceptance of the indwelling catheter and willingness to take part in the study

Exclusion Criteria:

-

Ages: 19 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females are only being recruited because this study looks at ovarian response
Enrollment: 5 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Urinary Pdg concentration | 4 months
  The primary endpoint of the study is luteal progesterone metabolite (pregnanediol; Pdg) excretion. Luteal Pdg will be compared in the pulsatile FSH cycle to the daily dose subcutaneous (SQ) cycle. Patients who conceive in the cycle of study will not have their conception cycle included in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Santoro, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pulsatile gonadotropin administration in in-vitro fertilisation — https://pubmed.ncbi.nlm.nih.gov/6144950/
- See also: Estradiol Priming Improves Gonadotrope Sensitivity and Pro-Inflammatory Cytokines in Obes — https://pubmed.ncbi.nlm.nih.gov/26425884/
- See also: Acute recapitulation of the hyperinsulinemia and hyperlipidemia characteristic of metabolic syndrome suppresses gonadotropins. — https://pubmed.ncbi.nlm.nih.gov/28158916/
- See also: Closed intravenous administration of gonadotropin-releasing hormone: safety of extended peripheral intravenous catheterization — https://pubmed.ncbi.nlm.nih.gov/2664612/
- See also: Effects of pulsatile intravenous follicle- stimulating hormone treatment on ovarian function in women with obesity. — https://pubmed.ncbi.nlm.nih.gov/37276947/
- See also: Pulsatile luteinizing hormone amplitude and progesterone metabolite excretion are reduced in obese women. — https://pubmed.ncbi.nlm.nih.gov/17440019/
- See also: Gonadotropin response to insulin and lipid infusion reproduces the reprometabolic syndrome of obesity in eumenorrheic lean women: a randomized crossover trial. — https://pubmed.ncbi.nlm.nih.gov/33838870/